CLINICAL TRIAL: NCT04592978
Title: Personalized Feedback Intervention to Address Hazardous Drinking and Alcohol-Opioid Interactions Among Adults With Chronic Pain.
Brief Title: Personalized Feedback Intervention for Alcohol and Opioid Use Among Adults With Chronic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Syracuse University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Joseph W. Ditre, Professor, Syracuse University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01AA028639 (NIH); R01AA028639 (NIH)
Record Dates: First submitted 2020-10-06; First posted 2020-10-19 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Alcohol Drinking; Pain; Opioid Use; Feedback, Psychological
Keywords: Alcohol; Opioids; Pain
MeSH Terms: conditions — Alcohol Drinking; Pain | interventions — Ethanol

STUDY DESIGN:
Intervention Model Description: Stage 1A will consist of 3 focus groups of 7 individuals used to develop and refine the pain-alcohol personalized feedback intervention (PFI).
  Stage 1B will employ a randomized controlled trial to compare the effects of the pain-alcohol PFI to a control PFI.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pain-Alcohol Personalized Feedback Intervention (Experimental)
  Interventions: Behavioral: Pain-Alcohol Personalized Feeback Intervention
- Control Personalized Feedback Intervention (Active Comparator)
  Interventions: Behavioral: Control Personalized Feedback Intervention

INTERVENTIONS:
Behavioral: Pain-Alcohol Personalized Feeback Intervention — The intervention will be designed to enhance knowledge regarding adverse pain-alcohol-opioid interrelations as well as increase motivation and intention to reduce hazardous drinking and positive attitudes and intentions regarding concurrent use of alcohol and prescription opioid medications.
  Arms: Pain-Alcohol Personalized Feedback Intervention
Behavioral: Control Personalized Feedback Intervention — The control intervention will incorporate personalized feedback relevant to exercise and nutrition but not address drinking reduction or pain-alcohol-opioid interrelations.
  Arms: Control Personalized Feedback Intervention

SUMMARY:
Over one-quarter of American adults engage in hazardous drinking (i.e., a pattern of alcohol consumption that increases risk for harmful consequences), which is the third leading cause of preventable death in the U.S. Rates of hazardous drinking are significantly higher among individuals with (vs. without) chronic pain. Moreover, 20% of individuals prescribed opioids endorse concurrent alcohol and opioid use, which may interfere with chronic pain treatment and lead to dangerous/potentially fatal health effects. No interventions to date have targeted either hazardous drinking or concurrent use of alcohol and opioids in the context of chronic pain. The current four-year R01 builds upon our past work by developing a brief, single-session, computer-based, personalized feedback intervention (PFI) designed to enhance knowledge regarding adverse pain-alcohol-opioid interrelations, increase motivation and intention to reduce hazardous drinking, and reduce positive attitudes and intention regarding concurrent use of alcohol and prescription opioid medications. Specifically, we will develop an integrated PFI for hazardous drinkers with chronic pain who are prescribed opioids (PA-PFI). Our approach will follow a staged model consistent with NIH guidelines for developing and standardizing behavioral interventions. Phase IA activities will involve collecting qualitative and quantitative feedback from three iterative focus groups (N = 21) to refine intervention content and evaluate treatment acceptability and feasibility. Phase IB activities will include a proof-of-concept and highly rigorous randomized clinical trial designed to compare PA-PFI to control PFI (C-PFI) among a sample of 174 hazardous drinkers with chronic pain who are currently prescribed opioid medications. This study represents an important and pivotal step in the larger landscape of translating basic research to more efficacious strategies for reducing hazardous drinking among underserved populations with medical comorbidities. This intervention would be highly disseminable and relevant to millions of hazardous drinkers with chronic pain. Given the collective public health impact of chronic pain, hazardous drinking, and concurrent alcohol-prescription opioid use, we believe the current study will yield findings that enhance scientific knowledge, enhance our understanding of mechanisms in reciprocal pain-alcohol-opioid relations, and inform the development of novel treatments for hazardous drinkers with chronic pain that are adaptable and easily implemented across a variety of healthcare settings.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 21 years of age
* Current hazardous drinker
* Current chronic pain
* Current use of prescription opioid medications.

Exclusion Criteria:

* Current alcohol or other substance use treatment
* Not being fluent in English
* Current psychiatric distress or thought disorder.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Actual)
Dates: Start 2021-07-30 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Change in knowledge of adverse pain-alcohol-opioid interrelations | Baseline and immediately after receiving the intervention
  Assessed via greater number of correct responses on the 10-item Pain Alcohol Opioid Knowledge Questionnaire (PAOKQ).
Change in motivation/readiness to reduce drinking | Baseline and immediately after receiving the intervention
  Assessed via Alcohol Ladder: a visual analogue contemplation ladder providing a single continuous metric of motivation and readiness to reduce drinking, where higher responses (range: 1-10) indicating greater motivation/readiness to change/reduce drinking.
Change in attitudes and intentions to co-use alcohol and opioids | Baseline and immediately after receiving the intervention
  Assessed via Alcohol-Opioid Co-Use Attitudes/Intentions (AOAI) measure, where greater scores (range: 16-62) indicate more positive attitudes and greater intentions to co-use alcohol and opioids.
Change in expectancies for pain-coping/reduction via drinking | Baseline and immediately after receiving the intervention
  Assessed via Expectancies for Alcohol Analgesia (EAA) measure, where greater EAA scores (range: 0-45) indicate greater expectancies for alcohol analgesia.
Change in hazardous drinking | Baseline and 3 month follow-up
  Assessed via scores on Alcohol Use Disorders Identification Test (AUDIT), where scores greater than or equal to 8 for males and 7 for females indicate the presence of hazardous drinking.
Change in frequency of alcohol-opioid co-use | Baseline and 3 month follow-up
  Assessed via self-reported number of days in which alcohol and prescription opioids were concurrently used in the past two weeks.

CONTACTS AND LOCATIONS:
Locations (1):
- Syracuse University, Syracuse, New York, United States

IPD SHARING:
Plan to Share IPD: No